CLINICAL TRIAL: NCT01872039
Title: A Multi-center, Randomized and Controlled Phase IV Study on the Efficacy and Safety of Two Dose Adjustment Regimens of Nicardipine Injection for Hypertensive Emergency
Brief Title: Post Marketing Study to Evaluate the Two Dose Regimens of Nicardipine Injection in Hypertensive Emergency Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACN-PD-2012001
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension Emergency; End-organ Damage
Keywords: Nicardipine; Hypertension; Calcium blocker
MeSH Terms: conditions — Hypertension | interventions — Nicardipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight-based adjustment group (Active Comparator): Dosage regimen according to the current Package Insert approved by SFDA
  Interventions: Drug: Perdipine injection
- Non-weight-based adjustment group (Experimental): Dosage regimen according to the Package Insert approved by FDA
  Interventions: Drug: Perdipine injection

INTERVENTIONS:
Drug: Perdipine injection — IV
  Other Names: nicardipine

SUMMARY:
To compare the efficacy and safety of two dose adjustment regimens (i.e. weight-based and non-weight-based) for the treatment of Chinese hypertensive emergency patients.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, open-label, randomized and controlled study. Subjects are selected from hypertensive emergency patients with a BP (Blood Pressure) of >180/120mmHg (SBP/DBP) and accompany with end target organ damage. All subjects are randomized into two groups receiving the Nicardipine Injection: Control Group (at a weight-based dose adjustment, i.e. according to the current Package Insert approved by SFDA) and Study Group (at a non-weight-based dose adjustment, i.e. according to the Package Insert approved by FDA).

Patients meet the inclusion/exclusion criteria are randomly allocated at 1:1 proportion to Control Group and Study Group. Before the treatment, investigators should define the target BP value for every subject according to different illness state, According to the BP, the dose of Nicardipine Injection is adjusted through different methods until reaching of target BP value. After reaching target BP value or 60min after the dosing initiation, BP and pulse rate are measured every 5~15min for 2h. Two to six hours after dosing, BP should be controlled at 160/100~110mmHg, and the maintenance dose is determined by the investigators according to the illness state.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure (SBP) ≥180mmHg and/or diastolic blood pressure (DBP) ≥120mmHg, and with the evidences or manifestations of end-organ damage (i.e. with any following hypertension emergency symptom: Chest pain, short breath, upper abdominal discomfort, syncope, vertigo, blurred vision, consciousness, hematuria or ischemic change under 12-lead ECG)
* Able to and voluntary to complete this study according to this study protocol, and sign the Informed Consent Form by himself/herself (or via his/her legal guardian)

Exclusion Criteria:

* Allergy to the Nicardipine Injection or its compositions
* Serious aortic valve stenosis
* Peri-operative hypertension
* Cerebral hemorrhage caused by the cerebrovascular malformation, hemangioma or cerebral infarction, cerebral hemorrhage into cerebral ventricle, and cerebral trauma with concomitant cerebral hemorrhage
* Other possible influencing factors for the safety or efficacy judgment in the investigators' opinions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with target BP | After 60 minutes of the treatment
  The target BP value is defined by investigators for every subject according to different illness state

SECONDARY OUTCOMES:
Blood pressure after the 6 hour treatment | At 6 hours
The time to get target BP | Within 2 hours after treatment
  The target BP value is defined by investigators for every subject according to different illness state
Safety assessed by the incidence of adverse events, vital signs and labo tests | For 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (5):
- China (5):
  - Beijing, Beijing Municipality
  - Shijiazhuang, Hebei
  - Harbin, Heilongjiang
  - Ürümqi, Xinjiang
  - Wuhan

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=ACN-PD-2012001